CLINICAL TRIAL: NCT00541112
Title: Phase II Multicenter Study of the Impact of the Therapeutic Sequence of Radiochemotherapy (50 Gy + Capecitabine + Oxaliplatin + Cetuximab) Followed by Total Mesorectal Excision Surgery Then Post-surgery Chemotherapy (FOLFOX 4 + Cetuximab) in Synchronous Locally Advanced or Metastatic Cancers of the Rectum With Metastases Resectable From the Start (T3-4 Nx or T2 N+ M1).
Brief Title: Radiation Therapy, Chemotherapy, and Cetuximab Followed by Surgery, Chemotherapy, and Cetuximab in Treating Patients With Locally Advanced or Metastatic Rectal Cancer That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity and lack of efficacy
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000565937; FRE-FNCLCC-ACCORD-14/0604 (Other: FNCLCC); EU-20759; 2006-003336-30 (EudraCT Number)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as capecitabine, oxaliplatin, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving radiation therapy together with combination chemotherapy and cetuximab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy and cetuximab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II clinical trial is studying how well giving radiation therapy together with chemotherapy and cetuximab followed by surgery, chemotherapy, and cetuximab works in treating patients with locally advanced or metastatic rectal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete remission rate at 6 months after neoadjuvant radiotherapy, capecitabine, and oxaliplatin (XELOX), and cetuximab followed by surgery, adjuvant FOLFOX 4, and cetuximab in patients with synchronous locally advanced or metastatic cancer of the rectum with resectable metastases (T3-4 Nx or T2 N+ M1).

Secondary

* Determine progression-free survival.
* Determine overall survival.
* Assess toxicities.
* Evaluate objective response in patients with measurable metastases.
* Determine the rate of local recurrence.
* Evaluate the downstaging and downsizing of patients with operable disease.
* Evaluate surgical complications in patients with operable disease.
* Evaluate biological markers predictive of response to cetuximab.

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy: Patients undergo radiotherapy for 5 weeks and receive concurrent oral capecitabine twice daily on days 1-5 of each week and oxaliplatin IV over 2 hours on day 1 of each week (XELOX). Patients also receive cetuximab IV on day 1 of the first week and on days 1-7 of weeks 2-5.
* Surgery: At 6 weeks after completing chemoradiotherapy, patients with resectable disease undergo surgery comprising total mesorectal excision. Patients with progressive disease, nonresectable tumor, or who require R2 surgery are removed from the study.
* Adjuvant therapy: Patients who undergo surgery, with or without removal of metastases, receive FOLFOX 4, comprising oxaliplatin IV over 2 hours, fluorouracil IV over 46 hours, and leucovorin calcium IV on day 1, and cetuximab IV. Treatment repeats every 2 weeks for up to 6 courses (approximately 3 months). Patients who have not undergone prior surgical resection of metastases may have surgery to remove metastases after completing this second regimen of chemotherapy.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Locally advanced (T3-4 Nx) or metastatic (T2 N+ M1) synchronous disease

    * Metastases must be resectable
  * Primary tumor examined by endorectal echography and MRI
* Measurable disease by thoraco-abdomino-pelvic scanner
* Disease considered susceptible to treatment with radiotherapy and chemotherapy
* No diffuse metastases considered nonresectable
* No acute occlusion not caused by colostomy

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* WBC ≥ 4,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 130 µmol/L
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients of must use effective contraception

Exclusion criteria:

* Contraindication to therapy with capecitabine, oxaliplatin, cetuximab, and/or radiotherapy
* Impossible to perform translational analyses
* Uncontrolled severe illness
* Severe renal or hepatic insufficiency
* Cardiac insufficiency or symptomatic coronary disease
* Sensitive peripheral neuropathy
* Uncontrolled diabetes
* Other malignancy within the past 10 years except previously treated basal cell skin cancer or carcinoma in situ of the cervix
* Impossible to participate in study due to geographic, social, or psychiatric reasons
* Patients who are under supervision or incarcerated

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior anticancer chemotherapy or radiotherapy for this cancer
* No therapy with coumarin anticoagulants, phenytoin, sorivudine, brivudine, antacids, or allopurinol
* No concurrent participation in another therapeutic study or receiving another experimental drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-10-29 (Actual); Primary Completion 2010-01-29 (Actual); Study Completion 2010-01-29 (Actual)

PRIMARY OUTCOMES:
Complete remission at ≥ 6 months by abdomino-pelvic-thoracic scan and a pelvic MRI

SECONDARY OUTCOMES:
Preoperative clinical response
Progression-free survival
Overall survival
Early toxicity before surgery
Early toxicity due to surgery (mortality at 30 days, postoperative complications, surgical recovery)
Late toxicity
Late radiotherapy toxicity by CTC AE v. 3.0
Objective response of measurable metastases by RECIST
Sexual function
Downstaging and downsizing of patients with operable disease
Surgical complications
Sphincter function
Predictive biomarkers of response to cetuximab

CONTACTS AND LOCATIONS:
Overall Officials: David Azria, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (10):
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif